CLINICAL TRIAL: NCT03144167
Title: Study of Prognostic Biomarkers of Survival at 6 Months for Patients Treated With Bevacizumab Glioblastomas in First Relapse After Failure of Radiochemotherapy
Acronym: SPECTROBEVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0027
Record Dates: First submitted 2017-04-27; First posted 2017-05-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients, aged 18-88, with glioblastoma (Other)
  Interventions: Other: Analysis of spectroscopic biomarkers of proliferation for six-month survival

INTERVENTIONS:
Other: Analysis of spectroscopic biomarkers of proliferation for six-month survival — Analysis of spectroscopic biomarkers of proliferation, glial reaction, infiltration and glutaminergic metabolism or glycolytic metabolism for six-month survival

SUMMARY:
No predictive factors are known for the response to the bevacizumab anti-angiogenic molecule (Avastin) given in the event of relapse of glioblastoma (GBM) following radiochemotherapy. Classical MRI with gadolinium injection and perfusion is not sufficient to predict survival and response or duration. We propose to evaluate the prognostic interest for 6-month survival of spectroscopic biomarkers of proliferation, glial reaction, infiltration and glutaminergic metabolism or glycolytic metabolism recorded at 7 and 28 days of application of the treatment.

These biomarkers are based on the increase of an index combining choline / Creatine (Cho / Cr), Glx / Cr (Glutamine and glutamate / Creatine), NAA / Cr (N acetyl aspartate / Creatine) and lactate / Cr ratios. The long-term objective is to predict the survival of these relapsed GBM patients at an early stage and to identify responder patients who would benefit from this expensive molecule and avoid using it in non-responding patients

ELIGIBILITY:
Inclusion Criteria:

* Patients, between 18 and 88 years, with glioblastoma (histologically proven) in first relapse after conventional treatment by surgery and temozolomide and radiotherapy
* Biological Criteria

  * Polymorphonuclear neutrophils> 1500 / mm3
  * Plates> 100,000 / mm3
  * SGOT-SGPT <5 at the upper limit of normal (ULN)
  * Bilirubin <1.5 x ULN
  * Creatinine <1.5 LSN and creatinine clearance
  * Proteinuria <1 g / 24 hours
  * Patient with health insurance
  * Consent signed by the patient if he is lucid, or failing that by the person of trust

Exclusion Criteria:

* Patients who can not benefit from bevacizumab for the following reasons:

  * Symptomatic cerebral or tumor hemorrhage
  * Karnofsky Index less than 50% or
* Patients already treated with an antiangiogenic molecule or Gliadel (diagnosis and recurrence).
* Coagulation disorders in case of injectable treatment (especially for avastin),
* Contraindications known to the MRI: Pace Makers, foreign bodies intraocular, electrodes ...
* Uncontrolled severe concomitant pathology, including another evolving cancer (with the exception of operative cutaneous tumors, in situ cancer of the cervix or breast treated).
* Uncontrolled Infection
* Uncontrolled hypertension (PAS> 160 mm Hg) despite optimized treatment
* Coronary artery disease or unstable arterial disease. Evolutionary aneurysm.
* Myocardial infarction dating from less than 6 months.
* Peripheral arterial or cerebrovascular accident occurring less than 6 months.
* Heart Failure> grade II NYHA
* Hemorrhagic Disease (Hemophilia, Willebrandt ...)
* Nephrotic syndrome with proteinuria> 2 g / 24 h
* History of haemoptysis dating less than 1 month.
* Pulmonary embolism dating less than 1 month.
* Surgical intervention (other than craniotomy or stereotactic biopsy) dating less than one month or essential and predictable surgery.
* History of digestive fistula or intestinal perforation with resolution less than 6 months.
* Hypersensitivity to bevacizumab or to any of the excipients mentioned in Composition.
* Hypersensitivity to Chinese hamster ovary (CHO) cells or to other human or humanized recombinant antibodies.
* Severe Myelosuppression
* Pregnant or nursing. Contraception should be prescribed if necessary during treatment.
* Persons deprived of liberty or placed under safeguard of justice (guardianship or curatorship),
* Subject involved in another search including an exclusion period still in progress at pre-inclusion
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Analyze 6-month survival defined as the time between inclusion in the protocol and death | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France